CLINICAL TRIAL: NCT01968421
Title: To Investigate the PRevention of OM-85 on Bronchiectasis Exacerbation (iPROBE): a Multicenter, Randomised, Double-dummy, Placebo-controlled Clinical Trial in Chinese Patients
Brief Title: Prevention of OM-85 on Bronchiectasis Exacerbation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University (Other); Capital Medical University (Other); Tianjin Medical University (Other); Zhejiang University (Other); China Medical University, China (Other); Tongji University (Other); Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Jinming Gao, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Bronchiectasis-Gao001; Vifro pharmaceuticals (Other Grant/Funding Number: PUMCHGao001)
Record Dates: First submitted 2013-10-17; First posted 2013-10-24 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Bronchiectasis With Acute Exacerbation
Keywords: OM-85, bronchiectasis, placebo, acute exacerbation
MeSH Terms: conditions — Bronchiectasis | interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OM-85 (Experimental): The subjects will be randomly received two courses of 7mg of OM-85 to take one oral capsule per day for 10 days a month for 3 consecutive months at the beginning of the study, then 3 months later with the same schedule for 1 year.
  Interventions: Drug: OM-85 BV
- Placebo (Placebo Comparator): The subjects will be randomly received two courses of 7mg of matching placebo to take one oral capsule per day for 10 days a month for 3 consecutive months at the beginning of the study, then 3 months later with the same schedule for 1 year.
  Interventions: Drug: OM-85 BV

INTERVENTIONS:
Drug: OM-85 BV — two courses of 7mg of OM-85 or matching placebo to take one oral capsule per day for 10 days a month for 3 consecutive months at the beginning of the study, then 3 months later with the same schedule for 1 year.
  Other Names: Bronchovaxom

SUMMARY:
Non-cystic fibrosis bronchiectasis is characterized by irreversible dilatation of the medium-sized bronchi as a result of airway injury due to recurrent or chronic inflammation and infection. Bronchiectasis airways are often colonized with bacterial species. Infections of the airways are thought to play an important role in bronchiectasis exacerbation. The non-specific prevention of recurrent airway infections by immunostimulating agents has gained growing scientific interest. OM-85, consisting extracts of eight kinds of bacteria important in respiratory infections, has shown the benefit for significantly reducing the incidence of exacerbations of chronic obstructive pulmonary disease (COPD). The purpose of this study is to investigate the PReventive effect of OM-85 on Bronchiectasis Exacerbation in Chinese patients (iPROBE).

This study is designed as a prospective randomised double-blind placebo-controlled multi-centred trial.

DETAILED DESCRIPTION:
Bronchiectasis is still a common chronic respiratory disease. Non-cystic fibrosis bronchiectasis is characterized by irreversible dilatation of the medium-sized bronchi as a result of airway injury due to recurrent or chronic inflammation and infection. Clinical features of bronchiectasis include chronic production of sputum often mucopurulent or purulent in nature, persistent bacterial colonization, recurrent lower respiratory tract infections. Bronchiectasis airways are often colonized with bacterial species. Infections of the airways are thought to play an important role in bronchiectasis exacerbation. Progressive lung damage in bronchiectasis results from a 'vicious cycle' of recurrent bacterial infection and a deregulated inflammatory response. The non-specific prevention of recurrent airway infections by immunostimulating agents has gained growing scientific interest. OM-85, consisting extracts of eight kinds of bacteria important in respiratory infections, has been known to support the respiratory tract resistance to the pathogens via activating pulmonary macrophages, increasing the ratio of CD4 to CD8 lymphocytes, and changing the level of a variety of cytokines in the lung. OM-85 has shown the benefit for significantly reducing the incidence of exacerbations of chronic obstructive pulmonary disease (COPD). Bronchiectasis exacerbations contribute substantially to rapid decline in lung function, reduced quality of life, and the medical costs. The purpose of this study is to investigate the PReventive effect of OM-85 on Bronchiectasis Exacerbation in Chinese patients (iPROBE).

This study is designed as a prospective randomised double-blind placebo-controlled multi-centred trial. A total of 244 patients with bronchiectasis, who have had at least one exacerbation of bronchiectasis in the previous year, will be included. The subjects will be randomly received two courses of 7mg of OM-85 or matching placebo to take one oral capsule per day for 10 days a month for 3 consecutive months at the beginning of the study, then 3 months later with the same schedule for 1 year.

We will investigate whether long-term therapy with an oral immunostimulant OM-85 can decrease exacerbations in patients with bronchiectasis over 1-year period. Besides, we will assess other outcomes including: the rate of event-based exacerbation, lung function parameters, the total scores on the St George's respiratory questionnaire and coughing, and inflammatory index. We hope that this study will provide novel information on the preventive effects of OM-85 treatment on bronchiectasis exacerbation and will address a knowledge gap for this poorly understood and under-studied disease.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the subject. The Informed Consent form will be signed.
* Subject/legal representative is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule or medication intake according to the judgment of the investigator.
* Subject with both genders is adult patients (>18 years) diagnosed with bronchiectasis by high-resolution computed tomography (HRCT) of chest within 3 years of study inclusion having had at least 1 acute exacerbation in the previous year when recruiting.

Exclusion Criteria:

* History of cystic fibrosis;
* Hypogammaglobulinaemia;
* Allergic bronchopulmonary aspergillosis;
* Active tuberculosis;
* Subject has been assigned to treatment in a study of the medication under investigation in this study in the previous 6 months.
* Subject has a history of chronic alcohol or drug abuse within the last 6 months.
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study.
* Subject has a known hypersensitivity to any components of OM85.
* Recent immunostimulant in last 3 months, cancer, stroke, severe cardiovascular disease, hepatic/kidney impairment, active TB, immuno-related diseases (RA and inflammatory bowel diseases), active ABPA.
* Subjects are free to withdraw from the study at any time, without prejudice to their continued care.
* Subject develops an illness that would interfere with his/her continued participation.
* Subject is noncompliant with the study procedures or medications in the opinion of the investigator.
* Subject takes prohibited concomitant medications as defined in this protocol (flu vaccine and pneumococcal vaccine).
* Subject withdraws his/her consent.
* There will have a confirmation of a pregnancy during the study, as evidenced by a positive pregnancy test.
* The sponsor or a regulatory agency requests withdrawal of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Gao, M.D., Principal Investigator — Peking Union Medical College Hospitak
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing
  - Shanghai Tongji University, Shanghai

REFERENCES:
- [Derived] Gao J, Gao X, Kong L. To investigate the prevention of OM-85 on bronchiectasis exacerbations (iPROBE) in Chinese patients: study protocol for a randomized controlled trial. Trials. 2014 Apr 29;15:150. doi: 10.1186/1745-6215-15-150. PMID 24773830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 1, 2015 was the starting date
Groups:
- OM-85: The subjects will be randomly received two courses of 7mg of OM-85 to take one oral capsule per day for 10 days a month for 3 consecutive months at the beginning of the study, then 3 months later with the same schedule for 1 year.
  OM-85: two courses of 7mg of OM-85 or matching placebo to take one oral capsule per day for 10 days a month for 3 consecutive months at the beginning of the study, then 3 months later with the same schedule for 1 year.
- Placebo: The subjects will be randomly received two courses of 7mg of matching placebo to take one oral capsule per day for 10 days a month for 3 consecutive months at the beginning of the study, then 3 months later with the same schedule for 1 year.
  OM-85: two courses of 7mg of OM-85 or matching placebo to take one oral capsule per day for 10 days a month for 3 consecutive months at the beginning of the study, then 3 months later with the same schedule for 1 year.
Period: Overall Study
Arm/Group | OM-85 | Placebo
Started | 99 (March 1, 2015 was the date for recruiting patients) | 97 (March 1, 2015 was the date for recruiting controls)
Starting Trial (starting to recuit first subject) | 99 | 97
Completed | 99 (Nov. 23, 2018 is the date for completing the trial) | 97 (Nov. 23, 2018 is the date for completing the trial)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 244 subjects were screened. 196 patients were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | OM-85 | Placebo | Total
Number analyzed (Participants) | 99 | 97 | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 70 | 145
  >=65 years | 24 | 27 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 57 | 110
  Male | 46 | 40 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 99 | 97 | 196
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — All subjects included in this trial were Chinese.
  Participants
    Race/Ethnicity | 99 | 97 | 196
Region of Enrollment [Number; unit: participants]
  China | 99 | 97 | 196

OUTCOME MEASURES:

1. Primary Outcome: Bronchiectasis Exacerbation
Description: the proportion of acute exacerbations
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: proportion of acute exacerbations
Arm/Group | OM-85 | Placebo
Number analyzed (Participants) | 99 | 97
proportion of acute exacerbations | 0.98 (1.19) | 0.75 (0.98)

2. Secondary Outcome: Life Quality
Description: (1)St George' s Respiratory Questionnaire (SGRQ); (2)Leicester Cough Questionnaire (LCQ)
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Lung Function
Description: Lung function parameters: FEV1, FVC, FEV1/FVC;
Time Frame: 1 year
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Rescue Medication
Description: Use of antibiotics and rapid-acting bronchodilator
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | OM-85 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/97
Serious Adverse Events (participants affected / at risk) | 2/99 | 1/97
Other Adverse Events (participants affected / at risk) | 4/99 | 7/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OM-85 (N=99) | Placebo (N=97)
Severe adverse events (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OM-85 (N=99) | Placebo (N=97)
Common cold (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT01968421/Prot_SAP_000.pdf